CLINICAL TRIAL: NCT02842385
Title: The Influence of Soft Tissue Thickness On Crestal Bone Changes Around Submerged and Nonsubmerged Implants: A Randomized Prospective Clinical Study
Brief Title: Soft Tissue Thickness on Submerged and Non Submerged Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Deniz Cengiz Özkaya, PhD, DDS, Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DCO-16
Record Dates: First submitted 2016-07-11; First posted 2016-07-22 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: Tooth Loss; Edentulousness
Keywords: soft tissue thickness; dental implant; crestal bone loss
MeSH Terms: conditions — Tooth Loss | interventions — Drug Implants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Nonsubmerged thick group (Active Comparator): Nonsubmerged type of implants placed with thick (>3 mm) soft tissue
  Interventions: Other: Implant
- Nonsubmerged thin group (Active Comparator): Nonsubmerged type of implants placed with thin (<3 mm) soft tissue
  Interventions: Other: Implant
- Submerged thick group (Active Comparator): Submerged type of implants placed with thick (>3 mm) soft tissue
  Interventions: Other: Implant
- Submerged thin group (Active Comparator): Submerged type of implants placed with thin (<3 mm) soft tissue
  Interventions: Other: Implant

INTERVENTIONS:
Other: Implant — One or two stages of implants within thin and thick gingiva were monitored 1.5 year after placement

SUMMARY:
Changes in the marginal bone level surrounding the implant are the frequently used parameters in assessing the short- and long-term success. Multiple biological and biomechanical factors have been reported to adversely affect marginal bone level. Recently, initial vertical mucosal tissue thickness has also been reported to have an impact on bone stability.The hypothesis of present study is that soft tissue thickness on implant placement has no positive impact of crestal bone remodeling.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the clinical and radiographical results of submerged and nonsubmerged implants with thin (<3 mm) and thick (>3 mm) soft tissue over 1.5 year after implant placement. All submerged and nonsubmerged implants were randomly placed as split-mouth. Clinical periodontal parameters were recorded. Crestal bone levels were analyzed from the day of implants inserted to 1.5 year after prosthetic loading on digitally standardized radiographs. Non-parametric test were used for statistically analysis.

ELIGIBILITY:
Inclusion Criteria:

* being older than 18 years of age
* generally healthy patients, no medical contraindication for implant surgery
* missing teeth in upper jaw posterior and more than one tooth in neighbourhood area
* no bone augmentation procedures before and during implant placement.

Exclusion Criteria:

* poor oral hygiene
* history of periodontitis
* smoking
* diabetes
* alcoholism
* taking medication which interferes soft and hard tissue healing
* bruxism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Crestal bone loss | Change from baseline crestal bone level at 4th month after placement,
  Crestal bone loss was measured on radiographs between baseline-4th month after placement
Crestal bone loss | Change from baseline crestal bone level at 6th month after placement,
  Crestal bone loss was measured on radiographs between baseline-6th month after placement
Crestal bone loss | Change from baseline crestal bone level at 12th month after placement,
  Crestal bone loss was measured on radiographs between baseline-12th month after placement
Crestal bone loss | Change from baseline crestal bone level at 18th month after placement,
  Crestal bone loss was measured on radiographs between baseline-18th month after placement

SECONDARY OUTCOMES:
Probing depth | Evaluation of probing depth at 4th month after placement (mm)
  Probing depth was measured with a plastic periodontal probe at 4th month after placement
Probing depth | Evaluation of probing depth at 6th month after placement (mm)
  Probing depth was measured with a plastic periodontal probe at 6th month after placement
Probing depth | Evaluation of probing depth at 12th month after placement (mm)
  Probing depth was measured with a plastic periodontal probe at 12th month after placement
Probing depth | Evaluation of probing depth at 18th month after placement (mm)
  Probing depth was measured with a plastic periodontal probe at 18th month after placement
Keratinized tissue level | Evaluation of keratinized tissue level at 4th month after placement (mm)
  Keratinized tissue level measured with a plastic periodontal probe at 4th month after placement
Keratinized tissue level | Evaluation of keratinized tissue level at 6th month after placement (mm)
  Keratinized tissue level measured with a plastic periodontal probe at 6th month after placement
Keratinized tissue level | Evaluation of keratinized tissue level at 12th month after placement (mm)
  Keratinized tissue level measured with a plastic periodontal probe at 12th month after placement
Keratinized tissue level | Evaluation of keratinized tissue level at 18th month after placement (mm)
  Keratinized tissue level measured with a plastic periodontal probe at 18th month after placement
Modified plaque index | Modified plaque index was recorded at 4th month after implant placement
  Modified plaque index was recorded at medial and distal surface of implants
Modified plaque index | Modified plaque index was recorded at 6th month after implant placement
  Modified plaque index was recorded at medial and distal surface of implants
Modified plaque index | Modified plaque index was recorded at 12th month after implant placement
  Modified plaque index was recorded at medial and distal surface of implants
Modified plaque index | Modified plaque index was recorded at 18th month after implant placement
  Modified plaque index was recorded at medial and distal surface of implants
Modified sulcus bleeding index | Modified sulcus bleeding index was recorded at 4th month after implant placement
  Modified sulcus bleeding index was recorded after 10 second of probing
Modified sulcus bleeding index | Modified sulcus bleeding index was recorded at 6th month after implant placement
  Modified sulcus bleeding index was recorded after 10 second of probing
Modified sulcus bleeding index | Modified sulcus bleeding index was recorded at 12th month after implant placement
  Modified sulcus bleeding index was recorded after 10 second of probing
Modified sulcus bleeding index | Modified sulcus bleeding index was recorded at 18th month after implant placement
  Modified sulcus bleeding index was recorded after 10 second of probing

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Cengiz Özkaya, PhD,DDS, Principal Investigator — Ege University, School of Dentistry

IPD SHARING:
Plan to Share IPD: Undecided